CLINICAL TRIAL: NCT03305458
Title: Improving Quality of Care in Child Mental Health Service Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH110620 (NIH)
Record Dates: First submitted 2017-10-04; First posted 2017-10-10 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Post Traumatic Stress Disorder; Technology; Child Abuse
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (Active Comparator): Trauma Focused Cognitive Behavioral Therapy
  Interventions: Behavioral: TFCBT
- Tablet-Facilitated TF-CBT (Experimental): Standard treatment with the addition of in-treatment/session iPad activities
  Interventions: Behavioral: eTFCBT

INTERVENTIONS:
Behavioral: TFCBT — treatment as usual
  Arms: Treatment as usual
Behavioral: eTFCBT — tablet-facilitated Trauma Focused Cognitive Behavioral Therapy (eTFCBT)
  Arms: Tablet-Facilitated TF-CBT

SUMMARY:
The investigators recently completed an NIMH R34 in which they piloted a patient- and provider-informed tablet-based toolkit designed to facilitate delivery of Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) - a treatment that was selected because it addresses a wide range of symptoms using techniques shared by other treatments for emotional and behavioral disorders. The tablet-based toolkit consists of numerous components (e.g., videos, interactive games, drawing applications) that are designed to facilitate provider-patient interactions in a way that enhances children's engagement and supports adherence to the treatment model. The tablet-based toolkit was very well received by children, caregivers, and providers in the pilot evaluation. Moreover, all benchmarks for feasibility were met or exceeded. This study proposes to conduct a hybrid effectiveness-implementation trial to examine the extent to which the tablet intervention may improve fidelity, engagement, and children's mental health outcomes. The investigators will conduct a randomized controlled trial with 120 mental health providers and 360 families in partnership with dozens of clinics in the Carolinas and Florida. Providers will be assigned randomly to tablet-facilitated vs. standard TF-CBT. Youth aged 8-16 years with clinically elevated symptoms of PTSD will be recruited. Baseline and 3-, 6-, 9-, and 12-month post-baseline assessments will be conducted by independent, blind evaluators. Sessions will be videorecorded for observational coding of engagement and fidelity by independent raters blind to study hypotheses. The investigators will also examine costs and conduct semi-structured interviews with families, providers, supervisors, and agency leaders to inform future dissemination and implementation initiatives. Technology-based resources that are scalable, easy to use, and designed for efficient integration into everyday practice may have sustained national impact.

DETAILED DESCRIPTION:
Assuring children access to the highest quality mental health care is a top national priority. Yet, quality of care continues to be highly variable in traditional service settings. Novel, scalable solutions are needed to address modifiable quality-of-care indicators in sustainable ways. To this end, provider fidelity and children's engagement are key correlates of clinical outcome and practical targets for intervention. There is tremendous opportunity to address both through technology. Studies in child education show that interactive games, touch-screen learning, and demonstration videos enhance engagement, knowledge, motivation, and learning. These benefits also may extend to the therapeutic context, where strategic integration of technology-based activities may enhance children's learning, strengthen the therapeutic alliance, and keep providers on protocol. The investigators recently completed an NIMH R34 in which they piloted a patient- and provider-informed tablet-based toolkit designed to facilitate delivery of Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) - a treatment that was selected because it addresses a wide range of symptoms using techniques shared by other treatments for emotional and behavioral disorders. The tablet-based toolkit consists of numerous components (e.g., videos, interactive games, drawing applications) that are designed to facilitate provider-patient interactions in a way that enhances children's engagement and supports adherence to the treatment model. The tablet-based toolkit was very well received by children, caregivers, and providers in the picot evaluation and all benchmarks for feasibility were met or exceeded. The investigators propose to conduct a hybrid effectiveness-implementation trial to examine the extent to which the tablet intervention may improve fidelity, engagement, and children's mental health outcomes. The investigators will conduct a randomized controlled trial with 120 mental health providers and 360 families in partnership with dozens of clinics in the Carolinas and Florida. Providers will be assigned randomly to tablet-facilitated vs. standard TF-CBT. Youth aged 8-16 years with clinically elevated symptoms of PTSD will be recruited. Baseline and 3-, 6-, 9-, and 12-month post-baseline assessments will be conducted by independent, blind evaluators. Sessions will be videorecorded for observational coding of engagement and fidelity by independent raters blind to study hypotheses. The investigators will also examine costs and conduct semi-structured interviews with families, providers, supervisors, and agency leaders to inform future dissemination and implementation initiatives. Technology-based resources that are scalable, easy to use, and designed for efficient integration into everyday practice may have sustained national impact.

ELIGIBILITY:
Inclusion Criteria:

* victim of at least one potentially traumatic event (e.g. sexual/physical assault, witnessed violence, disaster, serious accident)
* have at least one symptom on each PTSD symptom cluster (re-experiencing, avoidance, hyperarousal)

Exclusion Criteria:

* exhibits psychotic symptoms (active hallucinations, delusions, impaired thought processes) by caregiver or child
* significant cognitive disabilities, developmental delays, or pervasive developmental disorder
* active suicidal or homicidal ideations
* no consistent caregiver available to participate

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 713 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-10-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Not Randomized: Enrolled Providers will be randomized as soon as a family they referred enrolled into the study. Families did not enroll into the study or provider did not send a referral
Period: Overall Study
Arm/Group | Treatment as Usual | Tablet-Facilitated TF-CBT | Not Randomized
Started | 273 (117 children were randomized, 108 caregivers were randomized, 48 providers were randomized) | 326 (142 participants are children. 130 participants being caregivers/ parents enrolled into the study. 54 are providers) | 128 (All 128 are providers who are not randomized)
Completed | 138 | 195 | 0
Not Completed | 135 | 131 | 128
Not completed — Withdrawal by Subject | 50 | 46 | 93
Not completed — Lost to Follow-up | 85 | 85 | 35

BASELINE CHARACTERISTICS:
Groups:
- Not Randomized: As per the protocol, enrolled Providers will be randomized as soon as their family referral was enrolled into the study. Unfortunately the families they referred never enrolled into the study, or enrolled providers did not send a referral.
- Total: Total of all reporting groups
Arm/Group | Treatment as Usual | Tablet-Facilitated TF-CBT | Not Randomized | Total
Number analyzed (Participants) | 273 | 326 | 128 | 727
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 117 | 141 | 0 | 258
  Between 18 and 65 years | 148 | 178 | 128 | 454
  >=65 years | 8 | 7 | 0 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.0 (2.38) | 11.4 (2.38) | 36 (8.32) | 11.7 (2.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 215 | 262 | 116 | 593
  Male | 58 | 64 | 12 | 134
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 48 | 16 | 102
  Not Hispanic or Latino | 234 | 276 | 112 | 622
  Unknown or Not Reported | 1 | 2 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 21 | 2 | 32
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 2 | 7 | 0 | 9
  Black or African American | 99 | 102 | 26 | 227
  White | 147 | 178 | 89 | 414
  More than one race | 7 | 11 | 4 | 22
  Unknown or Not Reported | 8 | 6 | 6 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 48 | 16 | 102
  Not Hispanic or Latino | 234 | 276 | 112 | 622
  Unknown | 1 | 2 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 273 | 326 | 128 | 727

OUTCOME MEASURES:

1. Primary Outcome: Child Involvement Ratings Scale (CIRS)
Description: Child engagement will be measured via coding of audiotaped sessions by independent, trained raters who are blind to study purpose and hypotheses. The Child Involvement Ratings Scale (CIRS) will be used to code child engagement. Ten "child involvement" items-6 positive, 4 negative- are rated for each session on a 6-point scale. The minimum total score will be 0 and the maximum score is 50. For the outcome, a single average value will be presented. The positive-involvement items emphasize the extent to which children initiate discussions, demonstrate enthusiasm, self-disclose, and demonstrate understanding. Negative-involvement items address withdrawal or avoidance in treatment. Coders provide ratings based on two 10-min segments of session audiotapes (beginning at min 10 and min 40). Screening was conducted on enrolled participants.
Time Frame: 3 Month Timeline
Population: Measure was used on enrolled participants (Children).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment as Usual | Tablet-Facilitated TF-CBT
Number analyzed (Participants) | 62 | 49
units on a scale | 1.95 (.69) | 2.01 (.70)
Statistical Analysis 1: Comparison: Treatment as Usual vs Tablet-Facilitated TF-CBT; Test type: Superiority; To determine if child and caregiver engagement is affected by overall SPARK use, a 2-level MLM (level-1 child, level-2 provider) will be used. Engagement scores will be calculated per child and caregiver participant. An aggregate engagement score will determine if there are differences across conditions (SPARK + TF CBT vs standard TF-CBT) while accounting for the nesting providers

2. Primary Outcome: Provider Treatment Fidelity (TPOCS)
Description: Fidelity to the TF-CBT protocol will be measured by independent, trained raters who are blind to the study purpose and hypotheses, coding audiotaped treatment sessions. The TF-CBT Version of the Therapy Process Observational Coding System for Child Psychotherapy (TF-CBT TPOCS-S), modified for the eTF-CBT condition, will be used to assess provider fidelity to each TF-CBT component. Two raters will review video-recorded treatment sessions, assessing the presence or absence of specific techniques and rating their extensiveness on a 6-point scale.
  The total score will range from a minimum of 0 to the maximum 78. The outcome will be presented as a single average value.
Time Frame: 3 Month Timeline
Population: Measure was used on enrolled Randomized Providers
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment as Usual | Tablet-Facilitated TF-CBT
Number analyzed (Participants) | 33 | 31
units on a scale | .50 (.21) | .43 (.24)
Statistical Analysis 1: Comparison: Treatment as Usual vs Tablet-Facilitated TF-CBT; Test type: Superiority; To determine if provider fidelity is affected by overall SPARK use, a 2-level MLM (level-1 child; level-2 provider) will be used. Fidelity will be measured by the TF-CBT TPOCS-S. Providers' overall use of the toolkit will be calculated per child participant and averaged across toolkit content. Fidelity scores will be calculated per child participant such that each provider will have three ratings. An aggregate fidelity score will determine if there are differences across conditions (SPARK + TF-CBT vs. standard TF-CBT) while accounting for the nesting of providers

3. Secondary Outcome: Center for Epidemiological Studies Depression Scale for Children (CES-DC)
Description: assesses the severity of depressive symptomatology in children. It is a 20-item self-report measure with possible scores ranging from 0-60. Each questions has a scaling score of 0-3. With 0 being the lowest value stating 'Not at all' and 3 being the highest value stating 'A lot'. Total score over 15 is indicative of significant levels of depressive symptoms, showing worse outcome.
Time Frame: Baseline, 3 Month, 6 Month, 9 Month, 12 Month
Population: We encountered several challenges in conducting this study. First, some enrolled participants (caregivers and children) requested to discontinue their participation. Second, we experienced a high rate of loss to follow-up due to changes in contact information, such as disconnected phone numbers or children moving to a different foster home.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual | Tablet-Facilitated TF-CBT
Number analyzed (Participants) | 117 | 142
score on a scale
  Baseline Timeline: number analyzed (Participants) | 110 | 138
  Baseline Timeline | 25.21 (12.32) | 23.61 (11.86)
  3 Month Timeline: number analyzed (Participants) | 86 | 123
  3 Month Timeline | 20.88 (11.44) | 20.66 (11.92)
  6 Month Timeline: number analyzed (Participants) | 78 | 106
  6 Month Timeline | 19.22 (9.88) | 18.91 (10.21)
  9 Month Timeline: number analyzed (Participants) | 66 | 94
  9 Month Timeline | 18.35 (9.35) | 19.33 (10.73)
  12 Month Timeline: number analyzed (Participants) | 61 | 88
  12 Month Timeline | 16 (10.02) | 18.76 (11.152)
Statistical Analysis 1: Comparison: Treatment as Usual vs Tablet-Facilitated TF-CBT; Test type: Superiority; Response to the intervention will be evaluated with a piecewise longitudinal MLM that contains an additional level corresponding to time. Level-1 will correspond to time, level-2 to child, and level-to provider

4. Secondary Outcome: Therapeutic Alliance Scale for Children (TASC)
Description: The Therapeutic Alliance Score for Children is a 12-item measure of the child's alliance with the therapist using a 4-pt scale. It has good internal consistency and interrupter reliability. Measuring therapeutic alliance is one of the most reliable ways to determine the strength of this bond, and it allows the therapist to identify how comfortable their client might be in sharing their thoughts, experiences, struggles and goals with them throughout care. This scale completed by the adolescent participant aged 12-18, and there is a parallel version for the therapist to complete. Each item is rated on a 4 point scale ranging with 0 being the lowest value 'not at all' to 3 the highest value 'very much'. The lowest possible total score being 0 and the highest possible score (total score) would be 36. The higher the total score represents better outcome showing the strength of the child and therapist bond.
Time Frame: 3 Month
Population: At this point of time number of participant analyzed did drop due to participants discontinuing from the study or were missed at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual | Tablet-Facilitated TF-CBT
Number analyzed (Participants) | 83 | 117
score on a scale | 21.27 (3.73) | 20.67 (3.34)
Statistical Analysis 1: Comparison: Treatment as Usual vs Tablet-Facilitated TF-CBT; Test type: Superiority; Response to the intervention will be evaluated with a piecewise longitudinal MLM that contains an additional level corresponding to time. Level-1 will correspond to time, level-2 to child, and level-3 to provider

5. Secondary Outcome: Child/Adolescent Satisfaction Questionnaire (CASQ).
Description: The Child/Adolescent Satisfaction Questionnaire is a 15-item instrument that assesses child satisfaction with mental health treatment. The last three questions are open ended questions that do not provide value (these will not be measured/scored). The first twelve questions have a scoring scale between 1-5, with 1 being the lowest value ('Very much False') and 5 being the highest value with ('Very much True'). The total minimum score is 12 and the maximum total score being 60. The higher the total score represents a better outcome. Screening was given to enrolled children.
Time Frame: 3 Month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual | Tablet-Facilitated TF-CBT
Number analyzed (Participants) | 83 | 117
score on a scale | 51.20 (8.01) | 50.91 (8.79)
Statistical Analysis 1: Comparison: Treatment as Usual vs Tablet-Facilitated TF-CBT; Test type: Superiority; [other analysis details as in outcome 4, analysis 1]

6. Secondary Outcome: The Shame Measure
Description: 4-item instrument that assesses feelings of shame following abuse. With a score ranging 0-2, 0 being the lowest value 'Not true' and 2 being the highest value 'Very true'. The lowest possible total score is 0 and the highest possible total score is 8. The higher the score meant a worse outcome. Screening completed by enrolled children.
Time Frame: Baseline, 3 Month, 6 Month, 9 Month, 12 Month
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual | Tablet-Facilitated TF-CBT
Number analyzed (Participants) | 117 | 142
score on a scale
  Baseline Timeline: number analyzed (Participants) | 111 | 138
  Baseline Timeline | 2.40 (2.23) | 2.08 (2.23)
  3 Month Timeline: number analyzed (Participants) | 86 | 123
  3 Month Timeline | 1.58 (1.77) | 1.54 (2.01)
  6 Month Timeline: number analyzed (Participants) | 77 | 106
  6 Month Timeline | 1.34 (1.77) | 1.34 (1.94)
  9 Month Timeline: number analyzed (Participants) | 66 | 94
  9 Month Timeline | 1.21 (1.60) | 1.07 (1.71)
  12 Month Timeline: number analyzed (Participants) | 61 | 88
  12 Month Timeline | 1.02 (1.81) | 1.14 (1.78)
Statistical Analysis 1: Comparison: Treatment as Usual vs Tablet-Facilitated TF-CBT; Test type: Superiority; [other analysis details as in outcome 4, analysis 1]

7. Secondary Outcome: The Child and Adolescent Trauma Screen (CATS) - Youth Version
Description: 35-item instrument that assesses exposure to traumatic events and all 20 Diagnostic and Statistical Manual of Mental Disorder- Fifth Edition, Symptoms of PTSD. 20 items are scored ranging total value of 0-60; the minimum total score being 0 and the maximum total score being 60. Values ranging between 0-3, with the lowest possible score of 0 being 'Not at All' and 3 being the highest with 'All the time.' The higher values represent a worst outcome. Screenings complete with enrolled children.
Time Frame: Baseline, 3 Month, 6 Month, 9 Month, 12 Month
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual | Tablet-Facilitated TF-CBT
Number analyzed (Participants) | 117 | 142
score on a scale
  Baseline Timeline: number analyzed (Participants) | 111 | 137
  Baseline Timeline | 21.50 (13.03) | 21.66 (13.59)
  3 Month Timeline: number analyzed (Participants) | 85 | 123
  3 Month Timeline | 16.33 (11.58) | 16.83 (13.50)
  6 Month Timeline: number analyzed (Participants) | 78 | 106
  6 Month Timeline | 13.74 (11.06) | 14.51 (11.95)
  9 Month Timeline: number analyzed (Participants) | 66 | 93
  9 Month Timeline | 13.09 (12.39) | 12.10 (11.97)
  12 Month Timeline: number analyzed (Participants) | 61 | 88
  12 Month Timeline | 10.57 (11.61) | 12.33 (11.26)
Statistical Analysis 1: Comparison: Treatment as Usual vs Tablet-Facilitated TF-CBT; Test type: Superiority; [other analysis details as in outcome 4, analysis 1]

8. Secondary Outcome: Caregiver Satisfaction Questionnaire (CSQ)
Description: The Caregiver Satisfaction Questionnaire is a 15-item instrument that assesses caregiver satisfaction with mental health treatment. The last three questions are open ended questions that do not provide value (these will not be measured/scored). The first twelve questions have a scoring scale between 1-5, with 1 being the lowest value ('Very much False') and 5 being the highest value with ('Very much True').The minimum total score being 12 and the maximum total scores being 60. The higher the score represents a better outcome. Assessment given to only enrolled parent/caregivers and children. Screening was completed by enrolled caregivers/parents.
Time Frame: 3 Month
Population: Caregiver completed these assessments for each of their children. There are a number of parents that completed this assessment multiple times for each of their children who were enrolled.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual | Tablet-Facilitated TF-CBT
Number analyzed (Participants) | 79 | 120
score on a scale | 52.46 (7.64) | 52.79 (8.67)
Statistical Analysis 1: Comparison: Treatment as Usual vs Tablet-Facilitated TF-CBT; Test type: Superiority; [other analysis details as in outcome 4, analysis 1]

9. Secondary Outcome: Working Alliance Inventory (WAI-short Form)
Description: The WAI is a 12-item measure of the parent-therapist alliance using a 7-point scale (never to always). Scoring ranging between 1-7, with 1 being the lowest ('Never') and 7 being the highest with ('Always'). Total scores ranging between 12-84. Screening was completed by enrolled caregivers/parents. Higher score indicate a better therapeutic alliance.
Time Frame: 3 Month Timeline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual | Tablet-Facilitated TF-CBT
Number analyzed (Participants) | 82 | 116
score on a scale | 51.4 (7.85) | 51.03 (8.73)
Statistical Analysis 1: Comparison: Treatment as Usual vs Tablet-Facilitated TF-CBT; Test type: Superiority; [other analysis details as in outcome 4, analysis 1]

10. Secondary Outcome: Brief Problems Monitor (BPM)
Description: The BPM is a 19-item measure of emotional and behavioral functioning in children. The BPM is well-validated and comparable to the lengthier Child Behavior Checklist. The values range from 0-2 with 0 being the lowest value of 'Not True' and 2 being the highest value of 'Very True'. The lowest possible total score is 0 and the total highest possible score being 38. The higher the total score the worse outcome. Screening was completed with enrolled caregivers/parents.
Time Frame: Baseline, 3 Month, 6 Month, 9 Month, 12 Month
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual | Tablet-Facilitated TF-CBT
Number analyzed (Participants) | 117 | 142
score on a scale
  Baseline Timeline: number analyzed (Participants) | 108 | 139
  Baseline Timeline | 14.5 (7.78) | 14.9 (7.62)
  3 Month Timeline: number analyzed (Participants) | 85 | 125
  3 Month Timeline | 12.1 (8.07) | 13.3 (8.48)
  6 Month Timeline: number analyzed (Participants) | 78 | 103
  6 Month Timeline | 10.6 (8.94) | 12.7 (8.74)
  9 Month Timeline: number analyzed (Participants) | 59 | 90
  9 Month Timeline | 11.0 (8.99) | 12.1 (9.00)
  12 Month Timeline: number analyzed (Participants) | 60 | 88
  12 Month Timeline | 9.8 (8.99) | 11.9 (7.97)
Statistical Analysis 1: Comparison: Treatment as Usual vs Tablet-Facilitated TF-CBT; Test type: Superiority; [other analysis details as in outcome 4, analysis 1]

11. Secondary Outcome: Center for Epidemiologic Studies Depression Scale (CESD-R).
Description: The Center for Epidemiologic Studies Depression Scale is a 20-item self-report scale of depression completed by the enrolled caregiver. It is widely used and demonstrates excellent psychometric properties. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms. A score equal to or above 15 indicates a person at risk for clinical depression. Enrolled caregivers had multiple children enrolled meaning that caregivers with multiple children were asked more than once for each time point.
Time Frame: baseline, 3, 6, 9, 12 months Timeline
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual | Tablet-Facilitated TF-CBT
Number analyzed (Participants) | 117 | 142
score on a scale
  Baseline: number analyzed (Participants) | 110 | 141
  Baseline | 17.94 (14.59) | 18.28 (13.25)
  3 Month Timeline: number analyzed (Participants) | 87 | 128
  3 Month Timeline | 14.77 (13.71) | 16.23 (12.61)
  6 Month Timeline: number analyzed (Participants) | 80 | 106
  6 Month Timeline | 12.94 (12.99) | 23.88 (86.44)
  9 Month Timeline: number analyzed (Participants) | 65 | 100
  9 Month Timeline | 14.6 (12.80) | 15.62 (13.87)
  12 Month Timeline: number analyzed (Participants) | 67 | 96
  12 Month Timeline | 12.66 (12.90) | 14.91 (13.49)
Statistical Analysis 1: Comparison: Treatment as Usual vs Tablet-Facilitated TF-CBT; Test type: Superiority; [other analysis details as in outcome 4, analysis 1]

12. Secondary Outcome: The Child and Adolescent Trauma Screen (CATS) - Caregiver Version
Description: 35-item parent version of the CATS-Youth. CATS are given to enrolled Caregivers. A total symptom score is calculated by summing up the raw scores of items 1-20 (possible range = 0-60). The lowest value score of 0 being 'Never' and the highest value of 3 'Almost Always.' We recommend to use a cut-off ≥ 21 as indication of a clinically relevant level of symptoms. The higher the score means a worse outcome. Screening completed by enrolled caregiver/parents. Enrolled caregivers had multiple children enrolled meaning that caregivers with multiple children were asked more than once for each time point.
Time Frame: Baseline, 3 Month, 6 Month, 9 Month, 12 Month
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual | Tablet-Facilitated TF-CBT
Number analyzed (Participants) | 117 | 142
score on a scale
  Baseline: number analyzed (Participants) | 113 | 142
  Baseline | 21.16 (12.64) | 20.27 (12.65)
  3 Month: number analyzed (Participants) | 86 | 128
  3 Month | 13.80 (11.43) | 16.70 (12.26)
  6 Month: number analyzed (Participants) | 78 | 106
  6 Month | 13.95 (12.57) | 13.85 (12.09)
  9 Month: number analyzed (Participants) | 63 | 94
  9 Month | 13.62 (13.92) | 13.80 (12.23)
  12 Month: number analyzed (Participants) | 63 | 91
  12 Month | 10.22 (12.37) | 12.92 (12.06)
Statistical Analysis 1: Comparison: Treatment as Usual vs Tablet-Facilitated TF-CBT; Test type: Superiority; [other analysis details as in outcome 4, analysis 1]

13. Secondary Outcome: The Alabama Parenting Questionnaire
Description: 42-item measure to assess parenting practices. 13 questions were pulled to be utilized in these assessments. Scoring ranges are from 1- 5: 1 being 'Never', 2 being 'Almost never', 3 being 'Sometimes, 4 being 'Often', and 5 being 'Always'. Total minimum score being 13 and the highest possible score being 65. The higher score means worse outcome. With Assessment was given to Enrolled Caregivers/parents. Enrolled caregivers had multiple children enrolled meaning that caregivers with multiple children were asked more than once for each time point.
Time Frame: Baseline, 3 Month, 6 Month, 9 Month, 12 Month
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual | Tablet-Facilitated TF-CBT
Number analyzed (Participants) | 117 | 142
score on a scale
  Baseline Timeline: number analyzed (Participants) | 112 | 141
  Baseline Timeline | 43.72 (6.12) | 44.37 (6.23)
  3 Month: number analyzed (Participants) | 87 | 128
  3 Month | 43.26 (5.27) | 45.18 (5.87)
  6 Month: number analyzed (Participants) | 77 | 106
  6 Month | 43.44 (4.80) | 44.39 (6.32)
  9 Month: number analyzed (Participants) | 63 | 94
  9 Month | 43.33 (6.82) | 44.31 (6.52)
  12 Month: number analyzed (Participants) | 62 | 91
  12 Month | 43.05 (6.48) | 43.54 (5.81)
Statistical Analysis 1: Comparison: Treatment as Usual vs Tablet-Facilitated TF-CBT; Test type: Superiority; [other analysis details as in outcome 4, analysis 1]

14. Secondary Outcome: The Kessler 6
Description: Widely used the Kessler 6 measure of general distress that is well-validated. Assessment was given to Enrolled Caregivers.There are 6 items that are asked and each value scores ranging 0-4, with 0 being 'none of the time' and 4 being 'All of the time". With minimum total score would be 0 and maximum score would be 24. According to the scoring criteria proposed by Kessler 6, persons with a score of 13 or greater are likely to be experiencing severe mental illness. The higher total score represented a worse outcome. Screening was completed by enrolled caregivers/parents. Enrolled caregivers had multiple children enrolled meaning that caregivers with multiple children were asked more than once for each time point.
Time Frame: Baseline, 3 Month, 6 Month, 9 Month, 12 Month
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual | Tablet-Facilitated TF-CBT
Number analyzed (Participants) | 117 | 142
score on a scale
  Baseline Timeline: number analyzed (Participants) | 111 | 141
  Baseline Timeline | 6.10 (5.49) | 6.33 (5.44)
  3 Month Timeline: number analyzed (Participants) | 87 | 128
  3 Month Timeline | 4.86 (4.94) | 5.48 (4.70)
  6 Month Timeline: number analyzed (Participants) | 80 | 106
  6 Month Timeline | 4.96 (5.26) | 5.42 (4.80)
  9 Month Timeline: number analyzed (Participants) | 64 | 100
  9 Month Timeline | 5.05 (4.92) | 5.60 (5.24)
  12 Month Time: number analyzed (Participants) | 67 | 96
  12 Month Time | 4.25 (4.84) | 5.40 (5.59)
Statistical Analysis 1: Comparison: Treatment as Usual vs Tablet-Facilitated TF-CBT; Test type: Superiority; [other analysis details as in outcome 4, analysis 1]

15. Secondary Outcome: Evidence-Based Practice Attitude Scale (EBPAS)
Description: 15 items, assessing providers' perceptions of appeal of Evidence-Based Therapy, openness to innovation, perceived divergence with usual care (alphas .59-.90; M=.77).Scoring ranges from 0-4, with 0 being the lowest value ('Not at all') and 4 being the highest value ('To a Very Great Extent'). With the minimum score being 0 and the maximum score being 60. The higher Evidence-Based Practice Attitude Scale total score indicating more global positive attitudes toward adoption of Evidence-Based Practice.The higher the value reprents a better outcome. This assessment was given to enrolled providers.
Time Frame: baseline, post baseline at 12 Months
Population: We encountered several challenges in conducting this study. First, some enrolled participants (enrolled providers) requested to discontinue their participation. Second, we experienced a high rate of loss to follow-up due to changes in contact information, such as disconnected phone numbers or no longer working with the agency/clinic
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment as Usual | Tablet-Facilitated TF-CBT | Not Randomized
Number analyzed (Participants) | 48 | 53 | 126
units on a scale
  Baseline | 38.35 (6.21) | 38.83 (6.14) | 36.16 (6.90)
  Post Baseline at 12 months: number analyzed (Participants) | 28 | 34 | 52
  Post Baseline at 12 months | 39.39 (7.28) | 36.91 (7.66) | 35.19 (6.99)
Statistical Analysis 1: Comparison: Treatment as Usual vs Tablet-Facilitated TF-CBT vs Not Randomized; Test type: Superiority; [other analysis details as in outcome 4, analysis 1]

16. Secondary Outcome: Knowledge of Behavioral Principles as Applied to Children
Description: Assess understanding of the application of behavioral principles to youth. With the minimum score of 0 and maximum score of 25. the higher values represent a better outcome. Internal consistency=.42-.84; sensitivity to change. Screening completed with Enrolled Providers.
Time Frame: Baseline, Post Baseline at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment as Usual | Tablet-Facilitated TF-CBT | Not Randomized
Number analyzed (Participants) | 48 | 53 | 126
Participants
  Baseline | 48 | 53 | 123
  Post Baseline at 12 months | 27 | 35 | 53
Statistical Analysis 1: Comparison: Treatment as Usual vs Tablet-Facilitated TF-CBT vs Not Randomized; Test type: Superiority; [other analysis details as in outcome 4, analysis 1]

17. Secondary Outcome: Acceptability, Appropriateness and Feasibility Measure (AIMIAMFIM)
Description: 12-item measure to monitor and evaluate implementation efforts. This measure has been shown to have solid psychometric properties. Scaling is ranged from 1 to 5, with 1 being the lowest value with ('Completely Disagree') and 5 being the highest value ('Completely Agree'). With the total possible score ranging 12-60. With the lowest possible total score being 12 and the highest possible score being 60. The higher the values represent a better outcome. The higher scores indicate greater acceptability, appropriateness, and feasibility. Screening completed with enrolled providers.
Time Frame: baseline, Post baseline at 12 months
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment as Usual | Tablet-Facilitated TF-CBT | Not Randomized
Number analyzed (Participants) | 48 | 53 | 117
units on a scale
  Baseline | 53.94 (6.64) | 55.66 (5.40) | 52.10 (6.22)
  Post Baseline at 12 months: number analyzed (Participants) | 27 | 35 | 53
  Post Baseline at 12 months | 44.26 (7.40) | 52.86 (6.96) | 47.19 (8.58)
Statistical Analysis 1: Comparison: Treatment as Usual vs Tablet-Facilitated TF-CBT vs Not Randomized; Test type: Superiority; [other analysis details as in outcome 4, analysis 1]

18. Secondary Outcome: Computer Assisted Therapy Attitudes Scale
Description: 8-item measure design to assess attitudes toward computer use in treatment. Scaling on each question ranges 1-5 with 1 being the lowest value ('Strongly Disagree') and 5 being the highest value ('Strongly Agree'). The minimum total score would be 8 and the maximum total score being 40. The higher the value represents a better outcome. Assessment given only to enrolled providers.
Time Frame: baseline, post baseline at 12 months
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment as Usual | Tablet-Facilitated TF-CBT | Not Randomized
Number analyzed (Participants) | 48 | 53 | 125
units on a scale
  Baseline | 21.90 (3.36) | 19.79 (3.26) | 21.13 (2.87)
  Post Baseline: number analyzed (Participants) | 38 | 53 | 52
  Post Baseline | 20.96 (3.09) | 18.97 (3.45) | 20.67 (2.90)
Statistical Analysis 1: Comparison: Treatment as Usual vs Tablet-Facilitated TF-CBT vs Not Randomized; Test type: Superiority; [other analysis details as in outcome 4, analysis 1]

19. Secondary Outcome: Organizational Readiness for Implementing Change
Description: 12-item measure designed to assess an organization's readiness to implement new policies, programs, and practices. With values ranging between 1-5, 1 being the lowest of 'Disagree' and 5 being the highest with 'Agree'. The total minimum score being 12 and total maximum number being 60. The higher values represent a better outcome. Lower scores represent less organizational readiness for implementing change; Higher scores represent a more favorable organizational readiness for implementing change
Time Frame: baseline, post baseline at 12 months
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment as Usual | Tablet-Facilitated TF-CBT | Not Randomized
Number analyzed (Participants) | 48 | 53 | 126
units on a scale
  Baseline | 53.29 (7.15) | 51.87 (8.13) | 20.37 (7.87)
  Post Baseline at 12 month: number analyzed (Participants) | 28 | 34 | 53
  Post Baseline at 12 month | 46.57 (9.75) | 48.65 (9.74) | 47.13 (11.25)
Statistical Analysis 1: Comparison: Treatment as Usual vs Tablet-Facilitated TF-CBT vs Not Randomized; Test type: Superiority; [other analysis details as in outcome 4, analysis 1]

20. Secondary Outcome: TF-CBT Organizational Support Measure
Description: 19-item instrument to assess a community mental health organization's activities related to the delivery of Trauma-Focused Cognitive-Behavioral Therapy (TF-CBT). With values ranging between 1-5. 1 being the lowest with ' Strongly Disagree' and 5 being the highest with 'strongly agree'. The total minimum scores being 19 and the total maximum total scores being 95. The higher values represent a better outcome. Screening given to enrolled providers.
Time Frame: baseline, post baseline at 12 month
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment as Usual | Tablet-Facilitated TF-CBT | Not Randomized
Number analyzed (Participants) | 48 | 53 | 126
units on a scale
  baseline: number analyzed (Participants) | 48 | 53 | 117
  baseline | 62.96 (4.89) | 61.75 (7.80) | 62.48 (6.41)
  post baseline at 12 month: number analyzed (Participants) | 27 | 35 | 46
  post baseline at 12 month | 63.63 (6.05) | 63.43 (8.32) | 61.02 (7.95)
Statistical Analysis 1: Comparison: Treatment as Usual vs Tablet-Facilitated TF-CBT vs Not Randomized; Test type: Superiority; [other analysis details as in outcome 4, analysis 1]

21. Secondary Outcome: Burnout Measure
Description: screener that assesses providers' feelings about their work, and their perceptions of how their co-workers feel about the work they do. Scorings will range from 4- 28. Scaling value between 1-7, with 1 being the lowest value of 'Never' and 7 with the highest value of 'everyday'. Higher scores will mean worse outcome. Screening complete by enrolled providers.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment as Usual | Tablet-Facilitated TF-CBT | Not Randomized
Number analyzed (Participants) | 27 | 31 | 87
units on a scale | 10.11 (4.14) | 10.12 (4.10) | 10.17 (4.22)
Statistical Analysis 1: Comparison: Treatment as Usual vs Tablet-Facilitated TF-CBT vs Not Randomized; Test type: Superiority; [other analysis details as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: 52 weeks, 1 year
Description: Adverse events were monitored and assessed by our clinical supervisors.
Groups:
- Not Randomized: Providers who are enrolled into the study but did not have a family enrolled.
Arm/Group | Treatment as Usual | Tablet-Facilitated TF-CBT | Not Randomized
All-Cause Mortality (participants affected / at risk) | 0/267 | 4/320 | 0/126
Serious Adverse Events (participants affected / at risk) | 2/267 | 4/320 | 0/126
Other Adverse Events (participants affected / at risk) | 15/267 | 21/320 | 0/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment as Usual (N=267) | Tablet-Facilitated TF-CBT (N=320) | Not Randomized (N=126)
Suicide Ideations (Investigations) | 1 (1) | 0 (0) | 0 (0) — During a postbaseline assessment, the child participant disclosed previous suicidal ideation (e.g., thoughts of death and dying). He did not have intent or plan to engage in self-harm behaviors.
Self Harm (Investigations) | 1 (1) | 0 (0) | 0 (0) — A study interviewer was conducting a 3-month follow-up clinical assessment per study protocol. During the assessment, the caregiver participant disclosed the child's previous self-harm ideation.
Caregiver Death (Investigations) | 0 (0) | 4 (4) | 0 (0) — Caregivers have passed away. The deaths were not affiliated with the clinical study.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment as Usual (N=267) | Tablet-Facilitated TF-CBT (N=320) | Not Randomized (N=126)
Suicide Ideation/ Self Harm (Investigations) | 7 (7) | 9 (9) | 0 (0) — Participants have disclosed having suicide ideation and or self harm.
Patient taken to a Inpatient Clinic (Psychiatric disorders) | 1 (1) | 6 (6) | 0 (0)
Informing Therapist (Investigations) | 4 (4) | 4 (4) | 0 (0)
DSS Reports (Investigations) | 3 (3) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT03305458/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT03305458/SAP_001.pdf